CLINICAL TRIAL: NCT01236937
Title: Respiration Gated Laser Guided CT Lung Nodule Biopsy
Acronym: GENCTBIOPSY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Haseem Ashraf, Gentofte University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Gentofte CT guided biopsy
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-05

CONDITIONS: Lung Cancer
Keywords: CT, lung nodule biopsy, Respiration Gated, Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bellows-based breath hold biopsy (Active Comparator): CT guided biopsy is preformed with the use a bellows-based breath
  Interventions: Device: Bellows-based breath hold device
- No Bellows-based breath hold. (No Intervention): CT guided biopsy is preformed without the use a bellows-based breath
  Interventions: Device: Bellows-based breath hold device

INTERVENTIONS:
Device: Bellows-based breath hold device — Bellows-Based breath hold monitoring system:
  The bellows-based breath hold system (IBC, Mayo Clinic Medical Devices, USA) contains of 2 elements; one belt which is strapped around the thorax of the patient and a voltage controlled light unit with 8 lights. Belt stretch from respiratory motion is converted into voltage readings and displayed on the light unit giving biofeedback as different lights are activated depending on the dept of the respiration. Patients are instructed to keep respiration constant at a certain dept during the second the guide needle is inserted by controlling their breath with the help of the light unit. The patient is given a brief introduction to the system as to how the lights get turned on and off due to respiration motion before the biopsy is preformed.

SUMMARY:
The primary outcome of this study is to investigate the accuracy of respiration gated laser guided CT lung nodule biopsy through a prospective randomized trial using a bellows-based breath hold monitoring system. Secondary outcome is the rate of complications using laser guided CT biopsy in general and with bellows-based breath hold monitoring system. The study has approval from the The Danish National Committee on Biomedical Research Ethics (ref no: H-4-2010-fsp 1).

ELIGIBILITY:
Inclusion Criteria:

Patients with indeterminate lung nodules referred from the department of pulmonary medicine at Gentofte Hospital, Denmark for a CT guided biopsy are considered for inclusion in this study. The biopsy was preformed as part of regular clinical work up of the patient at the department of Radiology Gentofte Hospital, Denmark. Both men and women were included and no age restrictions were applied.

Exclusion Criteria:

Excluded from biopsy were those with poor pulmonary function test with a forced expired volume in the first second (FEV1) < 0.5 L, INR>1.2, blood cloth level under 200* and ECG with sign of ischemic heart disease. The trial is planned to begin 1.March 2010 and run for 2 years ending at 29 February 2012. During this time approx. 400 participants planned for biopsy are accepted to be included in the trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-03 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Accuracy of respiration gated laser guided CT lung nodule biopsy | After 2 years
  The primary outcome of this study is to investigate the accuracy of respiration gated laser guided CT lung nodule biopsy through a prospective randomized trial using a bellows-based breath hold monitoring system.

CONTACTS AND LOCATIONS:
Overall Officials: Haseem Ashraf, MD, PhD, Principal Investigator — Gentofte University Hospital, Department of Radiology; Paul Clementsen, MD, PhD, Study Chair — Gentofte University Hospital, Department of Pulmonology; Annete Nørgaard, MD, PhD, Study Chair — Gentofte University Hospital, Department of Pulmonology; Peter S. Myschetzky, MD, Study Chair — Gentofte University Hospital, Department of Radiology; Asger Dirksen, MD, PhD, Study Chair — Gentofte University Hospital, Department of Pulmonology; Zaigham Saghir, MD, Study Chair — Gentofte University Hospital, Department of Pulmonology
Locations (1):
- Gentofte University Hospital, Department of Radiology, Hellerup, Copenhagen, Denmark